CLINICAL TRIAL: NCT03846804
Title: Plasma-Based Next-Generation Sequencing for Pathogen Detection and Quantification in Children With Musculoskeletal Infections
Brief Title: Next-Generation Sequencing for Pathogen Detection and Quantification in Children With Musculoskeletal Infections
Acronym: KDG-002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Karius, Inc. (Industry)
Responsible Party: Principal Investigator, Jack Schneider, Assistant Professor of Clinical Medicine and Clinical Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1901296571
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Musculoskeletal Infection; Acute Hematogenous Osteomyelitis; Septic Arthritis; Osteomyelitis; Pyomyositis
Keywords: infection; plasma based next generation sequencing; blood culture; tissue culture; joint fluid culture; pathogen identification
MeSH Terms: conditions — Arthritis, Infectious; Osteomyelitis; Pyomyositis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Karius Test (Experimental): Participants will have additional blood drawn for the purposes of analysis with the Karius test.
  Interventions: Diagnostic Test: Karius Test

INTERVENTIONS:
Diagnostic Test: Karius Test — Next-generation sequencing of blood and synovial fluid samples for pathogen identification in children with musculoskeletal infections

SUMMARY:
The purpose of this study is to evaluate the use of a blood test: Karius® plasma-based next-generation sequencing test (Karius Test), to see if we can detect and measure the infection causing agent in children with musculoskeletal infections (MSKI).

DETAILED DESCRIPTION:
children admitted to Riley Hospital for Children (RHC) with musculoskeletal infections (osteomyelitis, septic arthritis, or pyomyositis) over a 12-month period will be prospectively enrolled. Eligible subjects will be identified by referral from the infectious diseases and orthopedic services at RHC. Blood samples will be obtained on the day of admission (within 48hrs), and 24 hours after the admission sample for real-time NGS (next-generation sequencing) testing at Karius Laboratory (Redwood City, CA). If a pathogen is identified by NGS, in either of the first two samples, subsequent samples will be sent every 48-72 hours while inpatient, and then collected every 1-2 weeks after hospital discharge, while being treated for MSKI (maximum 3 follow-up samples). If both of the initial inpatient NGS samples are negative, no further samples will be sent for NGS. Pathogen identification by NGS will be compared to standard cultures methods, and quantitative cfDNA (cell-free DNA) will be evaluated over time.

ELIGIBILITY:
Inclusion Criteria:

1. 6 months (to ensure adequate blood volume drawn) to 18 years of age.
2. Strong clinical suspicion of MSKI as evidenced by fever, osteoarticular pain (e.g. tenderness to palpation of a joint, bone pain, or refusal to bear weight); and elevated ESR (erythrocyte sedimentation rate) or CRP (C-reactive protein).

Exclusion Criteria:

* Subjects will be excluded if they have clinical evidence suggesting an alternative diagnosis; inability or unwillingness to consent for the study

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack G Schneider, MD, Principal Investigator — Indiana University School of Medicine - Pediatrics
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric Musculoskeletal Infections: Children 6 months to 18 years of age admitted to Riley Hospital for Children (Indianapolis, IN), from July 2019 to May 2022. Potential study participants were identified by daily screening of the pediatric infectious diseases and hospitalist patient censuses, and approached for enrollment if there was a strong clinical suspicion of MSKI as evidenced by fever, musculoskeletal pain (e.g. tenderness to palpation of a joint/bone, or refusal to bear weight); and elevated C-reactive protein (CRP) or erythrocyte sedimentation rate (ESR)
Period: Overall Study
Arm/Group | Pediatric Musculoskeletal Infections
Started | 38
Completed | 36
Not Completed | 2
Not completed — Refused blood draw | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Children with musculoskeletal infections
Arm/Group | Pediatric Musculoskeletal Infections
Number analyzed (Participants) | 36
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 7 [4 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 28
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Pathogen Identified by the Initial Karius Test (IP1) and Standard Culture Methods
Description: We evaluated the total number of participants that had a pathogen identified by the initial (IP1) Karius Test ("positive Karius Test").
  We compared the results of the Karius Test to cultures (gold standard) for each participant. Karius Test results that matched cultures results (same genus and species) were considered "positive agreement".
  We also evaluated at the number of participants who had negative cultures, but had a positive Karius Test.
Time Frame: Inpatient Sample 1 (IP1) - Within 48 hours of admission
Population: 36 children had a culture obtained (either blood or surgical or both) 33 children had a Karius Test available for analysis (1 sample failed quality control and 2 participants did not have an initial inpatient Karius Test sample drawn) 23 children had a positive culture, however, 1 participant with a positive culture had a Karius sample that failed quality control, leaving 22 available for positive agreement analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Musculoskeletal Infections
Number analyzed (Participants) | 36
Participants
  Children with Positive Culture (blood or surgical) | 23
  Children with a positive Karius Test (IP1): number analyzed (Participants) | 33
  Children with a positive Karius Test (IP1) | 26
  Positive agreement between culture and Karius Test (both tests identified the same organism): number analyzed (Participants) | 22
  Positive agreement between culture and Karius Test (both tests identified the same organism) | 15

2. Primary Outcome: Number of Participants With a Pathogen Identified by the Karius Test (at Time Point IP2) and Standard Culture Methods
Description: We evaluated the total number of participants that had a pathogen identified by the Karius Test ("positive Karius Test") at time point IP2 (within 48 hours of the initial sample).
  We compared the results of the Karius Test to those with a positive culture (gold standard) for each participant.
  Karius Test results that matched cultures results (same genus and species) were considered "positive agreement".
  Karius Test results that identified an organism different from the organism identified in culture were considered "discordant results" Karius Tests results that did not identify any organism were consider "negative"
Time Frame: Inpatient Sample 2 (IP2) - Within 48 hours of the initial sample
Population: 23 children had a positive culture, however, 5 participant with a positive culture did not have an IP2 Karius sample drawn, leaving 18 available for positive agreement analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Karius Test
Number analyzed (Participants) | 18
Participants
  Karius Test positive agreement with culture (blood or surgical) | 10
  Karius test discordant with culture (any) | 3
  Karius test negative | 5

3. Secondary Outcome: Microbial Cell Free DNA Level (cfDNA) in Molecules Per Microliter (MPM)
Description: We compared the microbial cfDNA level (on initial samples, IP1) between patients with non-severe MSKI to those with severe MSKI (defined as need for intensive care unit (ICU) care; infection in two or more non-contiguous anatomic sites (disseminated disease); need for more than 1 debridement procedure; deep vein thrombosis or thromboembolic disease; or pathologic fracture).
  Only those with a positive agreement between initial Karius Test (IP1) and culture were analyzed (n=15).
  Mann-Whitney U was used to compare median microbial cfDNA between those with non-severe vs. severe MSKI.
Time Frame: From hospital admission to hospital discharge, up to 3 months
Population: Patients with a positive agreement between the Karius Test and cultures
Measure: Median (Inter-Quartile Range); unit: MPM
Arm/Group | Karius Test
Number analyzed (Participants) | 15
MPM
  Severe Infection | 408 [358 to 49185]
  Non-Severe Infection | 322 [92 to 1357]
Statistical Analysis 1: Comparison: Karius Test; Test type: Other; p = 0.36, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Microbial Cell Free DNA (cfDNA) in Molecules Per Microliter (MPM) at Time Point IP1
Description: We evaluated whether cfDNA level (in MPM) correlated with C-reactive protein (CRP), erythrocyte sedimentation rate (ESR) and white blood cell count (WBC), common inflammatory markers followed in children with MSKI.
  Spearman's correlation was used to compare the MPM value to the CRP, ESR and WBC
Time Frame: Inpatient Sample 1 (IP1) - Within 48 hours of admission
Population: Patients with a positive agreement between Karius Test and culture who had a Karius Test, CRP, ESR and WBC obtained at time point IP1
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Karius Test
Number analyzed (Participants) | 15
Spearman's correlation coefficient
  MPM vs. CRP | 0.43
  MPM vs. ESR | 0.36
  MPM vs. WBC | 0.33

5. Secondary Outcome: Microbial Cell Free DNA (cfDNA) in Molecules Per Microliter (MPM) at Time Point IP2
Description: We evaluated whether cfDNA level (in MPM) correlated with C-reactive protein (a common inflammatory marker used to track inflammation in children with MSKI).
  Spearman's correlation was used to compare the MPM value to the CRP
Time Frame: Inpatient Sample 2 (IP2) - Within 48 hours of the admission sample
Population: Patients with a positive agreement between Karius Test and culture who had both a Karius Test and CRP obtained at time point IP2
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Karius Test
Number analyzed (Participants) | 7
Spearman's correlation coefficient | 0.79

6. Secondary Outcome: Microbial Cell Free DNA (cfDNA) in Molecules Per Microliter (MPM) at Timepoint IP3
Description: We evaluated whether cfDNA level (in MPM) correlated with C-reactive protein (a common inflammatory marker used to track inflammation in children with MSKI) at time point IP3 in participants with positive agreement between the Karius Test and culture.
  Spearman's correlation was used to compare the MPM value to the CRP
Time Frame: Inpatient Sample 3 (IP3) - Within 48 hours of the second inpatient sample
Population: Patients with a positive agreement between Karius Test and culture who had both a Karius Test and CRP obtained at timepoint IP3
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Karius Test
Number analyzed (Participants) | 3
Spearman's correlation coefficient | 1.0

7. Secondary Outcome: Microbial Cell Free DNA (cfDNA) in Molecules Per Microliter (MPM) at Time Point IP4
Description: We evaluated whether cfDNA level (in MPM) correlated with C-reactive protein (a common inflammatory marker used to track inflammation in children with MSKI).
Time Frame: Inpatient Sample 4 (IP4) - Within 48 hours of the third inpatient sample
Population: Patients with a positive agreement between Karius Test and culture who had both a Karius Test and CRP obtained at timepoint IP4
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Karius Test
Number analyzed (Participants) | 2
Spearman's correlation coefficient | NA — Only 2 participants with positive agreement between the Karius Test and culture had a sample drawn at time point IP4. Analysis requires at least 3 participants.

8. Secondary Outcome: Microbial Cell Free DNA (cfDNA) in Molecules Per Microliter (MPM) at Time Point OP1
Description: as for outcome 7
Time Frame: Outpatient Sample 1 (OP1) - 1-2 weeks after hospital discharge
Population: Participants with a Karius Test and CRP drawn at time point OP1
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Karius Test
Number analyzed (Participants) | 1
Spearman's correlation coefficient | NA — Only 1 participant with a positive agreement between the Karius Test and culture had an OP1 drawn. Analysis could not be done with only 1 participant

9. Secondary Outcome: Microbial Cell Free DNA (cfDNA) in Molecules Per Microliter (MPM) at Time Point OP2
Description: as for outcome 7
Time Frame: Outpatient Sample 2 (OP2) - 3-6 weeks after hospital discharge
Population: Participants with a Karius Test and CRP drawn at time point OP2
Measure: Number; unit: Spearman's correlation coefficient
Arm/Group | Karius Test
Number analyzed (Participants) | 1
Spearman's correlation coefficient | NA — Only 1 participant with a positive Karius Test drawn at OP2. Analysis could not be done with only 1 participant

10. Secondary Outcome: Microbial Cell Free DNA (cfDNA) in Molecules Per Microliter (MPM) at Time Point OP3
Description: as for outcome 7
Time Frame: Outpatient Sample 3 (OP3) - 6-8 weeks after hospital discharge
Population: Participants with a Karius Test and CRP drawn at time point OP3
Arm/Group | Karius Test
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through hospital follow up- up to 1 year
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Karius Test
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

LIMITATIONS AND CAVEATS:
The number of participants with the data for the secondary outcomes was very small, thus all of the secondary outcomes were underpowered to show a statistical difference. For secondary outcomes 7,8, and 9, there was not enough data to do the analyses. For secondary outcome 10, no patient data was collected because no patients followed up at this time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT03846804/Prot_SAP_000.pdf